CLINICAL TRIAL: NCT07095946
Title: Comparing the Effectiveness of the Intraligament Anesthesia Technique With the Inferior Alveolar Nerve Block Technique Using the Electronic Syringe in Children: A Random Clinical Study
Brief Title: Effectiveness of Intraligament vs IANB Anesthesia in Children Using Electronic Syringe
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tishreen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PED-DENT-Tishreen-University
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-05

CONDITIONS: Effectiveness of Anesthesia Using Electronic Syringe in Children in the Context of Endotopy Treatment
Keywords: Pediatric Dental Anesthesia Pulpitis Pain Management in Pediatric Dentistry Primary Teeth Endodontic Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electronic Syringe - IANB Technique (Experimental): Children receive inferior alveolar nerve block (IANB) using an electronic syringe. The injection is performed with controlled speed and pressure to ensure efficient pulpal anesthesia with minimal discomfort.
  Interventions: Device: Electronic syringe IANB Technique
- Electronic Syringe - Intraligamentary Technique (Experimental): Children receive intraligamentary anesthesia using an electronic syringe. The anesthetic is administered around the tooth ligament to provide localized anesthesia with minimal invasiveness and reduced discomfort.
  Interventions: Device: Electronic Syringe Intraligament Technique

INTERVENTIONS:
Device: Electronic Syringe Intraligament Technique — Use of an electronic syringe device to deliver local anesthesia using the periodontal ligament (PDL) technique in pediatric dental patients
  Arms: Electronic Syringe - Intraligamentary Technique
Device: Electronic syringe IANB Technique — Use of an electronic syringe device to deliver local anesthesia via the Inferior Alveolar Nerve Block Technique in pediatric dental patients
  Arms: Electronic Syringe - IANB Technique

SUMMARY:
This randomized clinical study aims to evaluate the efficacy and pain response of two local anesthesia techniques in pediatric dental treatment using an electronic syringe: ligament anesthesia and inferior alveolar nerve block (IANB). The study applies both techniques to the same sample, where each child undergoes pulpectomy for two different teeth, each under the influence of a different anesthesia technique, during two separate visits.

This study comes in the context of technological advancements in dentistry, which led to the development of computerized syringes as an alternative to traditional syringes. These devices are characterized by precise control of the anesthetic flow rate, as well as containing musical and auditory systems aimed at distracting the child and reducing feelings of fear and anxiety associated with dental treatment. Additionally, computerized syringes provide audible indicators showing the amount of anesthetic injected and support multiple injection modes such as rapid injection, slow injection, and ligament injection, allowing for more efficient and comfortable anesthetic delivery.

Pain intensity will be assessed during three stages of the treatment procedure: during anesthesia administration, during placement of the rubber dam, and during opening of the pulp chambers. Post-procedure pain will also be evaluated using an age-appropriate validated pain scale, along with assessing the satisfaction level of both the children and their parents regarding the use of the electronic syringe as an alternative anesthesia tool. These combined measures aim to provide a comprehensive understanding of the child's experience during dental treatment and contribute to improving anesthesia practices in pediatric dentistry.

ELIGIBILITY:
Inclusion Criteria:

* Cooperative children based on Frankl Behavior Rating Scale (Positive or Definitely Positive)
* No clinical signs or symptoms indicating irreversible pulpitis
* No periodontal ligament inflammation of the tooth to be treated
* Children aged between 5 and 9 years
* Children without systemic health problems

Exclusion Criteria:

* Children who are uncooperative based on Frankl Behavior Rating Scale (Negative or Definitely Negative)
* Presence of spontaneous or nocturnal pain
* Clinical signs and symptoms indicating irreversible pulpitis
* Presence of periodontal ligament inflammation of the treated tooth
* Child age older than 10 years or younger than 3 years
* Children with systemic health problems

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-05-28 (Actual); Primary Completion 2025-09-20 (Actual); Study Completion 2026-01-20 (Estimated)

PRIMARY OUTCOMES:
Success rate of electronic syringe anesthesia in pediatric dental procedures | During procedure (From the start of ligation anesthesia (30 seconds) and block anesthesia (3 to 5 minutes) until reaching the stage of pulp chamber opening)
Success rate of anesthesia technique | During procedure (From the start of ligation anesthesia (30 seconds) and block anesthesia (3 to 5 minutes) until reaching the stage of pulp chamber opening.)

CONTACTS AND LOCATIONS:
Overall Officials: Abdul Wahab Nourallah, Prof.Dr, Study Chair — Faculty of Pediatric Dentistry,Tishreen university
Locations (1):
- Faculty of Pediatric Dentistry, Tishreen University, Latakia, Latakia Governorate, Syria

IPD SHARING:
Plan to Share IPD: No
To protect the privacy of pediatric patients.